CLINICAL TRIAL: NCT04711941
Title: Effectiveness of a Novel Theory of Mind Training for People With Multiple Sclerosis: a Randomised Controlled Trial.
Brief Title: A ToM Training for People With Multiple Sclerosis: an Efficacy Study.
Acronym: ToM
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fondazione Don Carlo Gnocchi Onlus (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 5_25/07/2019
Record Dates: First submitted 2020-12-27; First posted 2021-01-15 (Actual); Last update posted 2021-05-06 (Actual); Status verified 2021-05

CONDITIONS: Multiple Sclerosis
Keywords: theory of mind; rehabilitation; multiple sclerosis; neurodegenerative disease
MeSH Terms: conditions — Multiple Sclerosis; Neurodegenerative Diseases

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ToM training (Experimental): ToM training was composed of six lessons two times a week. Through several types of stimuli, the trainer worked together with the participant to comprehend and hypothesize interpretations of the emotions and social interactions, providing discussion occasions to enhance the attribution of mental states and emotions. Every lesson had a duration of 45/60 minutes in order to avoid excessive fatigue in the participant.
  Interventions: Behavioral: Rehabilitation training
- Non mentalistic training (Active Comparator): ToM training was composed of six lessons two times a week. Through several types of stimuli, the trainer worked together with the participant to provide a historical and descriptive overview of cinema movies, TV news, documentaries, newspapers, and advertising. Every lesson had a duration of 45/60 minutes in order to avoid excessive fatigue in the participant.
  Interventions: Behavioral: Rehabilitation training

INTERVENTIONS:
Behavioral: Rehabilitation training — Rehabilitation with behavioural stimuli

SUMMARY:
Theory of Mind (ToM) is the ability to understand and attribute mental states to ourselves and others. People with Multiple Sclerosis (pwMS) could present an impairment of this ability, with negative consequences on their social relationships and Quality of Life (QoL). We aimed to design and implement a novel ToM rehabilitation training, testing its efficacy on the promotion of emotional and mental states understanding, on QoL and on the alexithymia traits.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of Relapsing-Remitting (RR), Secondary Progressive (SP) and Primary Progressive (PP) MS;
* age ≥ 18 and ≤ 75 years;
* years of education ≥ 5;
* no change of pharmacological treatment in the 6 months before the enrollment;
* no clinical relapses or use of steroid treatment during 3 months before the enrollment;
* provided informed consent for study participation.

Exclusion Criteria:

* history of nervous system disorders different from MS;
* unstable psychiatric illness, such as psychosis or major depression;
* severe disability with Expanded Disability Status Scale (EDSS) score > 7.5;
* severe cognitive impairment that would not enable PwMS to answer to questionnaires correctly (i.e. dementia), according to the patient's medical records.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2021-02-01 (Actual); Primary Completion 2021-05 (Estimated); Study Completion 2021-09 (Estimated)

PRIMARY OUTCOMES:
Reading the Mind from the Eyes (RMET) | 4 weeks
  A measure of affective ToM
Strange Stories | 4 weeks
  A measure of advanced ToM
Faux pas | 4 weeks
  A measure of both cognitive and affective advanced ToM
False Belief Task | 4 weeks
  A measure of cognitiveToM

SECONDARY OUTCOMES:
Toronto Alexithymia Scale (TAS-20) | 4 weeks
  A measure of Alexithymia traits
Multiple Sclerosis Quality of Life 54 questionnaire (MSQOL54) | 4 weeks
  A measure of Quality of Life in Multiple Sclerosis
Montreal Cognitive Assessment (MoCA) | 4 weeks
  A measure of global cognitive level
The Brief Repeatable Battery of Neuropsychological Test (BRB-NT) | 4 weeks
  A measure of cognitive functions in Multiple Sclerosis

CONTACTS AND LOCATIONS:
Locations (1):
- IRCCS Fondazione Don Carlo Gnocchi, Milan, Italy